CLINICAL TRIAL: NCT01494246
Title: Effectiveness of an E-mail Tracking Intervention Among the Continued Abstinence of Tobacco Consumption (TABATIC). A Randomized Controlled Multicentric Trial
Brief Title: Effectiveness of an E-mail Tracking Intervention Among the Continued Abstinence of Tobacco Consumption
Acronym: TABATIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other); Public Health Service of Cataluña (Other); Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PI11/00817
Record Dates: First submitted 2011-11-30; First posted 2011-12-16 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Tobacco Dependence; Cessation of Smoking
Keywords: Adult; computer-assisted instruction; electronic mail; program evaluation; smoking cessation/methods; continued abstinence
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electronic mail (Experimental)
  Interventions: Other: electronic mail
- brief advise (No Intervention)

INTERVENTIONS:
Other: electronic mail — Some e-mail will be sent to participants who will be in the intervention group in order to intensify the brief advise received for stop smoking.
  Other Names: e-mail, electronic mail, computer intervention,
  Arms: electronic mail

SUMMARY:
Objectives. To evaluate the effectiveness and cost effectiveness of clinical practice guide based intervention with two face-to-face visits and e-mail tracking compared to brief advice to obtain continued smoking abstinence at 6 and 12 months after intervention.

Methodology. simple randomized controlled multicentric trial. All smokers (N=1064) aged 18 or older that attend by any reason to the primary care center and that have an e-mail account and they checked it at least once a week will be invited to participate. The enrolled participants will be randomly divided into control (N=532) and intervention group (N=532). An intensive intervention, based on the recommendations of the clinical practice guides, that will include six contacts (2 face-to-face and 4 by e-mail) will be applied to the intervention group. Control group will receive brief advice.

The main dependent variable will be continued abstinence of tobacco consumption at six and twelve months after the beginning of the intervention which will be validated by and a carbon monoxide breathe analysis measured by a cooximeter in standard conditions. Secondary variables will include: stage change on the quitting smoking process and evaluation of the effectiveness on the reduction of the number of smoked cigarettes at six and twelve months after intervention. A descriptive analysis of all variables will be done. A multivariate analysis will be undertaken to assess differences among intervention and control group; logistic regression for dichotomic variables and lineal regression for continuous variables.

DETAILED DESCRIPTION:
In preliminary phase is planned to carry out 2 descriptive sub-studies: a qualitative one, which will reflect the views of patients and physicians regarding the use of email as a smoking cessation intervention, and another smoker's profile in relation to Information and Communication Technologies (ICT), which collects information on the actual use of them in smokers. The result of both will help to release data on the type of participants who would be involved in the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Smokers over 18 years old with an e-mail account who use frequently. (Smoker is an individual who smokes any amount of tobacco, whatever this amount it is.
* E-mail regular user is the one who uses it as a way of communication at least once per week)

Exclusion Criteria:

* Not regular e-mail users,
* patients who have diseases that advise not to stop smoking:
* Terminal diseases
* Serious psychiatric disorders
* Active addiction to other psychoactive drugs
* Patients in smoking cessation process
* whatever the cause that does not allow to understand goals and methodology of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1064 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in smoking status and maintenance in smoking cessation | the outcome measure is studied at 6 and 12 months
  The term used to name long term abstinence over 6 months is continuous abstinence.

SECONDARY OUTCOMES:
point prevalence abstinence | the outcome measure is studied at 3, 6 and 12 months
  In case ok not reaching abstinence, will be measured if a subject has changed of stage in "transtheoretical model of Prochaska and DiClemente".
self-reported tobacco consumption | the outcome measure is studied at 3, 6 and 12 months
self-reported smoking reduction | the outcome measure will be studied at 3, 6 and 12 months
  In case not reaching abstinence
stage of change in Prochaska cycle | the outcome measure will be studied at 3,6 and 12 months
used time by professionals to achieve patients stop smoking | the outcome measure will be studied at 3, 6 and 12 months
used time by participants | the outcome measure will be studied at 3, 6 and 12 months
cost to get smoking help in primary care service | the outcome measure will be studied at 3, 6 and 12 months
  The estimated cost of helping people to leave smoking in regular conditions

CONTACTS AND LOCATIONS:
Overall Officials: José L Ballvé Moreno, MD, Study Chair — Institut Català de la Salut; Marc Casajuana, Economist, Study Chair — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina; Lourdes Clemente, MD, Study Chair — Servicio Aragones De Salud; Laura Díaz Gete, MD, Principal Investigator — Institut Català de la Salut; Elena M Briones Carrió, Statistician, Study Chair — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina; Mireia Fàbregas Escurriola, MD, Study Chair — Institut Català de la Salut; Elisa Puigdomènech Puig, Byologist, Study Chair — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina; José L del Val, MD, Study Chair — Institut Català de la Salut; Soraya Fernández Maestre, nurse, Study Chair — Institut Català de la Salut; Carlos Martín Cantera, MD, Ph D, Study Chair — Institut Català de la Salut. Research Unit of Barcelona, IDIAP Jordi Gol. Department of Medicine, University Autonomus of Barcelona; Ricardo Almon, MD, PhD, Study Chair — Family Medicine Research centre School of Health and medical Sciences. Örebro University
Locations (1):
- Jordi Gol i Gurina Foundation. Research Unit of Barcelona. Lifestyles Research Group., Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Diaz-Gete L, Puigdomenech E, Briones EM, Fabregas-Escurriola M, Fernandez S, Del Val JL, Ballve JL, Casajuana M, Sanchez-Fondevila J, Clemente L, Castano C, Martin-Cantera C; Grupo Estudio TABATIC. Effectiveness of an intensive E-mail based intervention in smoking cessation (TABATIC study): study protocol for a randomized controlled trial. BMC Public Health. 2013 Apr 18;13:364. doi: 10.1186/1471-2458-13-364. PMID 23597262